CLINICAL TRIAL: NCT03630939
Title: A Multicenter, Double-Blind, Randomized, Vehicle-Controlled Phase 1/2a Study to Evaluate the Safety, Pharmacokinetics, and Efficacy of Topical ESR-114 Gel in Subjects With Plaque Psoriasis
Brief Title: A Study to Evaluate the Safety, Pharmacokinetics, and Efficacy of Topical ESR-114 in Subjects With Plaque Psoriasis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Escalier Biosciences B.V. (Industry)
Collaborators: Innovaderm Research Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ESR-114-101
Record Dates: First submitted 2018-08-10; First posted 2018-08-15 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Psoriatic Plaque

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- ESR-114 1.5% (Experimental): ESR-114 1.5% Topical Gel BID for 6 weeks
  Interventions: Drug: ESR-114
- ESR-114 5.0% (Experimental): ESR-114 5.0% Topical Gel BID for 6 weeks
  Interventions: Drug: ESR-114
- Vehicle Gel (Placebo Comparator): Placebo Topical Gel BID for 6 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: ESR-114 — ESR-114 Topical Gel
  Arms: ESR-114 1.5%; ESR-114 5.0%
Other: Placebo — Placebo Topical Gel
  Arms: Vehicle Gel

SUMMARY:
This is a multicenter, double-blind, randomized, vehicle-controlled, parallel-group proof-of-concept study designed to assess the safety, tolerability, pharmacokinetics, and preliminary efficacy of topically applied ESR-114 following twice daily (BID) application for 42 days (6 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Subject has a history of plaque psoriasis for at least 6 months.
* Subject has PGA of mild (2) or moderate (3) at Day 1.
* Subject has total LSS of ≥6 at Day 1.
* Subjects with plaque psoriasis-affected BSA to be treated of 1% to 15% at Screening and Day 1.

Exclusion Criteria:

* Subject has non-plaque psoriasis at Screening and Day 1.
* Subject has a history of skin disease or presence of skin condition that, in the opinion of the Investigator, would interfere with the study assessments at Screening and Day 1.
* Subject has used any topical therapy to treat psoriasis within 2 weeks prior to Day 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2018-08-09 (Actual); Primary Completion 2019-06-05 (Actual); Study Completion 2019-06-12 (Actual)

PRIMARY OUTCOMES:
Change in Total Lesion Severity Score | 6 weeks
  Change from Baseline in Total Lesion Severity Score (sum of scores for Induration, Erythema, & Desquamation; score range: 0-12; lower score is better outcome) at Week 6

SECONDARY OUTCOMES:
Proportion of subjects with clear or almost clear on the Physician Global Assessment | 6 weeks
  Proportion of subjects with clear or almost clear on the Physician Global Assessment (PGA) at Week 6
Proportion of subjects with PASI75 | 6 weeks
  Proportion of subjects with PASI75 at Week 6
Change from Baseline in erythema score over time | 6 weeks
  Change from Baseline in erythema score (score range: 0-4; lower score is better outcome) at Weeks 1, 2, 4, and 6
Change from Baseline in induration score over time | 6 weeks
  Change from Baseline in induration score (score range: 0-4; lower score is better outcome) at Weeks 1, 2, 4, and 6
Change from Baseline in desquamation score over time | 6 weeks
  Change from Baseline in desquamation score (score range: 0-4; lower score is better outcome) at Weeks 1, 2, 4, and 6

CONTACTS AND LOCATIONS:
Overall Officials: Allison Luo, MD, Study Chair — Escalier Biosciences B.V.
Locations (10):
- United States (8):
  - Study Site 19, Santa Monica, California
  - Study Site 16, Tampa, Florida
  - Study Site 17, Fridley, Minnesota
  - Study Site 14, Raleigh, North Carolina
  - Study Site 12, Austin, Texas
  - Study Site 11, College Station, Texas
  - Study Site 15, Houston, Texas
  - Study Site 18, San Antonio, Texas
- Canada (2):
  - Study Site 13, Peterborough, Ontario
  - Study Site 10, Montreal, Quebec